CLINICAL TRIAL: NCT05188183
Title: Pragmatic Trial of Remote tDCS and Somatosensory Training for Phantom Limb Pain With Machine Learning to Predict Treatment Response
Acronym: PLP-EVEREST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003323
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- M1 anodal home-based tDCS and somatosensory training (Experimental): Investigators will use the Soterix Medical 1X1 tDCS mini-CT stimulator device (© Soterix Medical Inc.) an home-based tDCS device used in several clinical trials with no adverse events. It sends a low-level current from the positive electrode, anode, to the negative electrode, cathode. During tDCS, low amplitude direct currents are applied via scalp electrodes and penetrate the skull to enter the brain. HB-TDCS will be combined with somatosensory training that will be performed during the self-administration of tDCS, including 20 sessions over 4 weeks.
  Interventions: Device: M1 anodal home-based tDCS; Behavioral: Somatosensory Training
- Usual Care (Experimental): Usual care includes pharmacological treatments, physical therapy, occupational therapy and/or behavioral therapy that the subject is receiving.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: M1 anodal home-based tDCS — During tDCS, low amplitude direct currents are applied via scalp electrodes and penetrate the skull to enter the brain. Direct current will be transferred by a saline-soaked pair of surface sponge electrodes (35 cm2) and delivered by a specially developed, battery-driven, constant current stimulator with a maximum output of 10 mA.
  Arms: M1 anodal home-based tDCS and somatosensory training
Behavioral: Somatosensory Training — The somatosensory training will be performed during the self-administration of tDCS, including 20 sessions over 4 weeks. Sessions will start with relaxation exercises using a body scan technique, whereby subjects in a relaxed state will be instructed to sequentially interchange their mind to different regions of the body while perceiving it and establishing contact with the body part. Subjects will be asked to concentrate on any feeling (kinetic, kinesthetic or exteroceptive) related to each body part. Phantom exercises will involve the use of imagined movements of the phantom limb. Therefore, patients will be asked to perform general exercises with their phantom limb. Exercises will include hip, knee, ankle, and toe movements.
  Arms: M1 anodal home-based tDCS and somatosensory training
Other: Usual Care — Usual care includes pharmacological treatments, physical therapy, occupational therapy and/or behavioral therapy that the subject is receiving.
  Arms: Usual Care

SUMMARY:
The investigators have designed a pragmatic trial of home-based transcranial direct current stimulation (tDCS) for phantom limb pain (PLP), the PLP-EVEREST trial (PLP-EffectiVEness pRagmatic Stimulation Trial) to test a portable device that would reach underrepresented populations and would validate this therapy in a more pragmatic setting. Subjects will be randomized to home-based tDCS of the primary motor cortex (M1) with somatosensory training or usual care only (including their current pharmacological treatments, physical therapy, and occupational therapy). The investigators will therefore test the effectiveness of home-based tDCS and somatosensory training in a real-world, home-based setting. The Investigator will compare patients randomized to this combined strategy vs. usual care alone (subjects from this group will be offered combined treatment at the end of the trial). The investigators hypothesize that the combined strategy will be associated with a significantly larger Cohen's d effect size (at least 1) compared to the control group.

DETAILED DESCRIPTION:
The investigators have designed a pragmatic trial of home-based tDCS for PLP, the PLP-EVEREST trial (PLP-EffectiVEness pRagmatic Stimulation Trial) to test a portable device that would reach underrepresented populations and would validate this therapy in a more pragmatic setting. Subjects will be randomized to home-based tDCS of the M1 with somatosensory training or usual care only (including their current pharmacological treatments, physical therapy, and occupational therapy). The investigators will therefore test the effectiveness of home-based tDCS and somatosensory training in a real-world, home-based setting. The investigator will compare patients randomized to this combined strategy vs. usual care alone (subjects from this group will be offered combined treatment at the end of the trial). The investigators hypothesize that the combined strategy will be associated with a significantly larger Cohen's d effect size (at least 1) compared to the control group.

The investigators will perform a pragmatic, parallel randomized clinical trial. Investigators will recruit 290 participants with upper and/or lower bilateral or unilateral limb amputation and phantom limb pain in the chronic phase. All participants will be randomized to receive 20 daily sessions (4 weeks) of active anodal M1 home-based tDCS combined with somatosensory training or usual care. The participants will participate in 23 visits over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age - older than 18 years
2. Limb amputation
3. Patients who experience PLP regularly (at least once a week)
4. Pain not attributable to other causes, such as peripheral inflammation
5. Current chronic pain as defined by an average pain of at least 4 on the numeric rating scale (NRS, 0: no pain, 10: worst imaginable pain)

Exclusion Criteria:

1. Any clinically significant or unstable medical or psychiatric disorder
2. History of substance abuse in the past 6 months (according to the DSM-V criteria for substance use disorder with six or more symptoms)
3. Uncompensated psychiatric disorder
4. Previous significant neurological history with current significant neurological deficits
5. Previous neurosurgical procedure with craniectomy that would affect current distribution of tDCS
6. Contraindications to tDCS (implanted brain medical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for Phantom Limb Pain | From Baseline to Visit 22 (at 4 weeks)
  The VAS is a common assessment that asks subjects to self-reportedly measure their pain on a visual scale (i.e., unbearable to none). Investigators will use the VAS to determine subjects' pain scores. Subjects will rate their pain from 0 - indicating no pain at all, to 10 - indicating the worst pain felt. This scale is also colored, from green (at 0) to red (at 10), as a visual indicator of pain. This assessment tool is frequently used in many research studies evaluating pain levels in phantom limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the trial and after publication of the primary manuscript, the investigators plan to publish the de-identified dataset following the guidelines of our institution (Spaulding Rehabilitation Hospital/Partners Healthcare and Harvard Medical School).